CLINICAL TRIAL: NCT05319951
Title: Effect of Different Liquids Intake in Vasovagal Reaction After Whole Blood Donation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou Blood Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Different liquids intake
Record Dates: First submitted 2020-12-01; First posted 2022-04-11 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Blood Donation
MeSH Terms: interventions — Water

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Oral Rehydration Salts Power (iii) (Experimental): Dissolve 2 packs of Oral Rehydration Salts Power (iii) (5.125g/pack) in 500ml water and let the subjects drink it up in 20 minutes prior to donation.
  Interventions: Drug: Oral Rehydration Salts power (iii)
- water with white granulated sugar (Experimental): Dissolve 2 packs of Taikoo white granulated sugar (5g/pack) in 500ml water and let the subjects drink it up in 20 minutes prior to donation.
  Interventions: Dietary Supplement: water with white granulated sugar
- recommended water intake (Placebo Comparator): Recommend the subjects to drink up 500ml water in 20 minutes prior to donation.
  Interventions: Dietary Supplement: water

INTERVENTIONS:
Drug: Oral Rehydration Salts power (iii) — Dissolve 2 packs of Oral Rehydration Salts Power (iii) (5.125g/pack) in 500ml water and let the subjects drink it up in 20 minutes prior to donation.
  Other Names: Sichuan Emeishan Pharmaceutical Co., Ltd. 20210402 5100621103491
  Arms: Oral Rehydration Salts Power (iii)
Dietary Supplement: water with white granulated sugar — Dissolve 2 packs of Taikoo white granulated sugar (5g/pack) in 500ml water and let the subjects drink it up in 20 minutes prior to donation.
  Arms: water with white granulated sugar
Dietary Supplement: water — Recommend the subjects to drink up 500ml water in 20 minutes prior to donation.
  Arms: recommended water intake

SUMMARY:
we compared the effect of 3 different kinds of liquids (water, Oral Rehydration Salt 3 and white granulated sugar water) intake in Vasovagal Reaction After Whole Blood Donation

DETAILED DESCRIPTION:
Vasovagal reaction is the most common type of blood donation reaction. The main cause of this reaction is the decrease of blood volume. Therefore, fluid supplement before blood donation has been proved to be effective in preventing the vagal reaction after blood donation. It was proved that isotonic (sugar & salt) drink intake before blood donation had a significant effect on reducing vasovagal reaction.

However, in 2002, WHO recommended the new reduced osmolarity rehydration formula with better taste. Oral Rehydration Salt 3 has been produced according to WHO formula with standard ingredient and easy to prepare. In addition, in Guangdong culture, sugar water is regarded as a tonic, more easily accepted. So, the aim of our study was to compare the effects of 500 ml water with Oral Rehydration Salt 3, white granulated sugar and conventional recommended water intake prior to blood donation on blood donation reaction after whole blood donation, in order to understand the effect of different liquid supplement on blood donation reaction and the willingness of blood donation again.

ELIGIBILITY:
Inclusion Criteria:All blood donors donated whole blood in Guangzhou Blood Center during study.

-

Exclusion Criteria:Blood donors who were deferral by blood screening result and other situations.

-

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6250 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2021-11-26 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
vasovagal reaction rate | 1-3days
  vasovagal reaction rate in three groups

SECONDARY OUTCOMES:
rate of willingness to donate blood again | 3days
  rate of willingness to donate blood again in three groups

CONTACTS AND LOCATIONS:
Overall Officials: Guiyun Xie, MPH, Study Chair — Guangzhou Blood Center; Jinyan Chen, MPH, Principal Investigator — Guangzhou Blood Center; Shijie Li, Study Director — Guangzhou Blood Center
Locations (1):
- Guangzhou Blood Center, Guangzhou, Guangdong, China